CLINICAL TRIAL: NCT05921877
Title: AMH May Not be a Good Index of Ovarian Reserve in Patients With Functional Hypothalamic Amenorrhea
Brief Title: AMH and Functional Hypothalamic Amenorrhea
Acronym: AMELIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5321
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Amenorrhea Secondary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with functional hypothalamic amenorrhea: Women aged 15-34 years Diagnosis of functional hypothalamic amenorrhea (for at least 2 years) No interventions to be administered
  Interventions: Diagnostic Test: venous sampling
- Healthy controls: Women aged 15-34 years Normal menstrual cycles No interventions to be administered
  Interventions: Diagnostic Test: venous sampling

INTERVENTIONS:
Diagnostic Test: venous sampling — venous sampling

SUMMARY:
The purpose of this study is to analyze AMH levels in patients with prolonged FHA (more than 2 years). Based on previous studies, we can assume that prolonged FHA may mimic a condition of primary hypogonadotropic hypogonadism, due to a lasting interruption of gonadotropin release. Furthermore, after the resumption of the spontaneous menstrual cycle, we will reanalyze AMH levels, which we hypothesize to find higher. If our hypotheses are confirmed correct, we could support the thesis that AMH is not a good index of ovarian reserve in patients with functional hypothalamic amenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 15-34 years.
* Diagnosis of functional hypothalamic amenorrhea (for at least 2 years).
* Signature of informed consent.

Exclusion Criteria:

* Polycystic ovary syndrome
* Taking oral contraceptives in the previous three months
* Other clinically relevant endocrinopathies
* positive MAP-test (Medroxyprogesterone acetate test)
* Estroprogestin replacement therapy
* Autoimmune disorders
* Failure to sign informed consent

Ages: 15 Years to 34 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Patients with functional hypotalamic amenorrhea (FHA) will be recruited from the DH of Dysfunctional Gynecology (UOSD Diagnostic and Medical Therapy of Menstrual Dysfunction and Marital Infertility) Department of Women's, Children's and Public Health Sciences of the A. Gemelli IRCCS University Polyclinic Foundation. Possible enrollment in the study protocol will not affect or alter in any way the patient's clinical course or adherence to good clinical practice guidelines. A group of healthy controls will also be enrolled, respecting the same exclusion criteria, from among the patients afferent to the Day Hospital of Dysfunctional Gynecology (healthy control is defined as: patient not suffering from functional hypothalamic amenorrhea, not from polycystic ovary syndrome and with 10-12 menstrual cycles per year).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-16 (Estimated); Primary Completion 2024-06-16 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
AMH assay | 12 months
  Check serological AMH levels in patients with FHA for at least 2 years and compare them with AMH levels in healthy women.

SECONDARY OUTCOMES:
To correlate AMH levels with other parameters | 12 months
  Correlate serologic AMH levels with antral follicle count (AFC). Verify serologic AMH levels in previously FHA patients after resumption of spontaneous menstruation, i.e., at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rosanna Apa, Rome, Italy

IPD SHARING:
Plan to Share IPD: No